CLINICAL TRIAL: NCT04494919
Title: Two Different Novel Stent Placement Technique for Intestinal Stenosis Assisted by an Ultrafine Endoscope
Brief Title: Novel Stent Placement Technique for Intestinal Stenosis Assisted by an Ultrafine Endoscope
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UFE-1.0
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrafine Endoscope Assisted: The self-expanding metal stent (SEMS) implantation was conducted using an ultrafine endoscope (UFE) (GIF-XP260NS; Olympus, Tokyo, Japan). The UFE researched the stricture, and a guidewire was inserted into the endoscopic working channel. The guidewire was left. And the endoscope was withdrawn. The normal colonoscope was exchanged under the reverse guidance of the guidewire. Finally, a metal, uncovered SEMS was placed along the guidewire.
  Interventions: Device: Ultrafine Endoscope

INTERVENTIONS:
Device: Ultrafine Endoscope — The reversal of the normal colonoscope (CV-260SL; Olympus, Tokyo, Japan) along the guidewire to replace the UFE (GIF-XP260NS; Olympus, Tokyo, Japan).

SUMMARY:
Colorectal cancer is the third most common cancer worldwide and results in 8-25% acute malignant bowel obstruction. Since Dohmoto et al. first applied and reported the self-expanding metal stents (SEMS) in the treatment of colorectal stenosis, they have been widely used not only as an alternative treatment as a bridge to surgery (BTS), but also as a mean of palliative option for stenosing lumen in clinical practice. Numerous publications have reported that the stent placement technique showed 75% to 100% technical success rates and 84% to 100% clinical success rates. However, it is sometimes difficult to place due to the distorted anatomy or acute angulations in patients and other conditions with poor endoscopic visualization with the normal colonoscope. The aims of this study were to present our results with two novel SEMS implantation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients with colorectal cancer stenosis
* Patients with intestinal stent implantation in digital subtraction angiography room

Exclusion Criteria:

* Patients undergoing conventional intestinal stent implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colorectal stricture underwent novel intestinal stent implantation methods assised by ultrafine endoscope.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The technical success rate | 1 hour
  the ratio between the patients with correctly placed SEMS and those scheduled for SEMS implantation.

SECONDARY OUTCOMES:
The clinical success rate | 24 hours
  the ratio between the patients with regressive signs and symptoms of obstruction (within 24 h) and those succeeded for SEMS implantation.
The adverse events rate | 2 year
  the ratio between the patients with adverse events (like perforation, bleeding, and reobstruction) and those succeeded for SEMS implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China